CLINICAL TRIAL: NCT05011877
Title: A Strategy to Improve Management and Prolong LIFe Without Readmission for hYpercapnic Patients: The Simplify Project
Brief Title: The Simplify Project
Acronym: SIMPLIFY
Status: Recruiting | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 21-103
Record Dates: First submitted 2021-07-20; First posted 2021-08-18 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Acute Hypercapnic Respiratory Failure
Keywords: Acute Hypercapnic Respiratory Failure; Patient Readmission; Mortality; Sleep Disorders, Intrinsic
MeSH Terms: conditions — Respiratory Insufficiency; Sleep Disorders, Intrinsic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute Hypercapnic Respiratory Failure patients with Sleep Disorders: Acute Hypercapnic Respiratory Failure patients with Sleep Disorders
  Interventions: Device: High-flow nasal cannula therapy
- Acute Hypercapnic Respiratory Failure patients without Sleep Disorders: Acute Hypercapnic Respiratory Failure patients without Sleep Disorders
  Interventions: Device: High-flow nasal cannula therapy

INTERVENTIONS:
Device: High-flow nasal cannula therapy — High-flow nasal cannula therapy (HFNC) (from 25 - 60 L/min based on patient's tolerance) will be used in 21 participants during one additional sleep study to investigate its acute impact on reducing sleep abnormalities. Inspired fraction of oxygen will be titrated to maintain patient SpO2 similar to the levels during standard oxygen therapy.

SUMMARY:
The high frequency of unplanned hospital visits of patients with chronic hypercapnic respiratory failure (e.g., chronic obstructive pulmonary disease, obesity-related hypoventilation) constitutes a major public health problem. Most patients admitted for acute exacerbations (AHRF) have additional comorbidities, especially sleep disorders. Often untreated, sleep disorders contribute to multiple readmissions (≈70% at one year) and increase readmission costs. The investigators will: 1) identify these patients early during unplanned hospital admissions and perform sleep studies using EEG and oximetry before hospital discharge and two months after to compare sleep abnormalities in the two moments; 2) investigate the association between sleep abnormalities in the two sleep studies with clinical outcomes (1-year readmission and death); 3) investigate the acute effects of high-flow nasal cannula (HFNC) to treat sleep abnormalities as a simplified alternative. The investigators anticipate sleep abnormalities during the hospital stay and two months after discharge will be associated with poor clinical outcomes (readmission, death) and HFNC to acutely reduce sleep abnormalities.

DETAILED DESCRIPTION:
The investigators will perform sleep studies using nocturnal EEG measurements and oximetry 1) while the participants are still in the hospital but have reached relative clinical stability (≥48 h after admission, not in ICU and pHv ≥7.36) and 2) two months after hospital discharge at the participant's home. Sleep studies will be performed from 5:00 pm to 8 am. EEG measurements will be performed using a portable monitor (Prodigy Sleep System, Cerebra, Winnipeg, Canada). Sleep assessment will be performed offline. The ORP will be continuously quantified and ORP-derived indices will be calculated. Nocturnal oximetry will be used for detecting sleep desaturation episodes. Comorbidities (e.g., obesity, diagnosed lung or heart disease, Charlson comorbidity index) and exacerbations/hospitalization in the previous year will be identified.

In 21 participants, the investigators will perform one additional sleep study with the participants breathing with high-flow nasal cannula therapy (HFNC) to investigate the acute impact (i.e., during one night) of HFNC on reducing sleep abnormalities. HFNC will be set from 25 - 60 L/min based on participant's tolerance and the inspired fraction of oxygen will be titrated to maintain patient SpO2 similar to the levels during standard oxygen therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients requiring an unplanned hospitalization or emergency room visit due to an acute hypercapnic respiratory failure exacerbation (AHRF), not on home noninvasive or invasive ventilation, neuromuscular disease (e.g., spinal cord injury) or central nervous system disorders (e.g., cerebral vascular accident, Alzheimer), absence of tracheotomy, and non-morbidly obese.

Exclusion Criteria:

* Patients with AHRF due to drug overdose
* Ventilatory support (noninvasive or invasive ventilation) is needed before or during the sleep studies or if an acute deterioration (e.g., cerebral vascular accident, cardiac arrest) happens before or during the sleep studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute hypercapnic respiratory failure (pH <7.35 and PaCO2 > 45 mmHg at admission) admitted for an unplanned hospitalization or emergency room visit.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
1-year hospital readmission and 1-year mortality | 1 year
  The primary endpoint is to compare the rate of 1-year Hospital readmission and mortality between patients with acute hypercapnic respiratory failure with vs. without sleep abnormalities during the home sleep study measured by the odds ratio product (ORP) and the 2017 American Academy of Sleep Medicine rules

SECONDARY OUTCOMES:
Hospital length of stay | Through study completion, an average of 1 year
  The secondary endpoint is to compare the length of stay during the hospital admission between patients with acute hypercapnic respiratory failure with vs. without sleep abnormalities during the sleep study performed at the hospital measured by the odds ratio product (ORP) and the 2017 American Academy of Sleep Medicine rules
Need of ventilatory support | Through study completion, an average of 1 year
  The secondary endpoint is to compare the need of invasive and non-invasive ventilatory support between patients with acute hypercapnic respiratory failure with vs. without sleep abnormalities during the sleep study performed at the hospital measured by the odds ratio product (ORP) and the 2017 American Academy of Sleep Medicine rules
Need of ICU admission | Through study completion, an average of 1 year
  The secondary endpoint is to compare the need of ICU admission between patients with acute hypercapnic respiratory failure with vs. without sleep abnormalities during the sleep study performed at the hospital measured by the odds ratio product (ORP) and the 2017 American Academy of Sleep Medicine rules
In-hospital mortality | Through study completion, an average of 1 year
  The secondary endpoint is to compare the rate of in-hospital mortality between patients with acute hypercapnic respiratory failure with vs. without sleep abnormalities during the sleep study performed at the hospital measured by the odds ratio product (ORP) and the 2017 American Academy of Sleep Medicine rules
HFNC effects on sleep depth according to the ORP range | 15 hours
  In 21 patients. Time spend in different ORP ranges during the sleep study which the patients used the standard oxygen therapy and the night which the patients used HFNC.
Sleep depth according to the ORP during the sleep study performed at the hospital and at home | 15 hours
  Time spend in different ORP ranges during the sleep study performed in the hospital vs. at home.
HFNC effects on sleep depth according to the AASM criteria | 15 hours
  In 21 patients. Time spend in different sleep stages (AASM 2017 rules) during the sleep study which the patients used the standard oxygen therapy and the night which the patients used HFNC.
HFNC effects on the prevalence of sleep abnormalities | 15 hours
  In 21 patients. The prevalence of sleep abnormalities during the sleep study which the patients used the standard oxygen therapy and the night which the patients used HFNC.
Sleep depth according to the AASM at the hospital vs. home | 15 hours
  Time spend in different sleep stages (AASM 2017 rules) during the sleep study performed at the hospital vs. at patient's home.
Prevalence of sleep abnormalities at the hospital vs. home | 15 hours
  The prevalence of sleep abnormalities during the sleep study performed at the hospital vs. at home.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Brochard, MD, PhD, Principal Investigator — Unity Health Toronto - St. Michael's Hospital
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Younes M, Ostrowski M, Soiferman M, Younes H, Younes M, Raneri J, Hanly P. Odds ratio product of sleep EEG as a continuous measure of sleep state. Sleep. 2015 Apr 1;38(4):641-54. doi: 10.5665/sleep.4588. PMID 25348125
- [Background] Sharma S, Mather PJ, Chowdhury A, Gupta S, Mukhtar U, Willes L, Whellan DJ, Malhotra A, Quan SF. Sleep Overnight Monitoring for Apnea in Patients Hospitalized with Heart Failure (SOMA-HF Study). J Clin Sleep Med. 2017 Oct 15;13(10):1185-1190. doi: 10.5664/jcsm.6768. PMID 28859720
- [Background] Younes M, Soiferman M, Thompson W, Giannouli E. Performance of a New Portable Wireless Sleep Monitor. J Clin Sleep Med. 2017 Feb 15;13(2):245-258. doi: 10.5664/jcsm.6456. PMID 27784419
- [Background] Berry RB, Brooks R, Gamaldo C, Harding SM, Lloyd RM, Quan SF, Troester MT, Vaughn BV. AASM Scoring Manual Updates for 2017 (Version 2.4). J Clin Sleep Med. 2017 May 15;13(5):665-666. doi: 10.5664/jcsm.6576. No abstract available. PMID 28416048
- [Background] Dres M, Younes M, Rittayamai N, Kendzerska T, Telias I, Grieco DL, Pham T, Junhasavasdikul D, Chau E, Mehta S, Wilcox ME, Leung R, Drouot X, Brochard L. Sleep and Pathological Wakefulness at the Time of Liberation from Mechanical Ventilation (SLEEWE). A Prospective Multicenter Physiological Study. Am J Respir Crit Care Med. 2019 May 1;199(9):1106-1115. doi: 10.1164/rccm.201811-2119OC. PMID 30818966
- [Background] Drouot X, Roche-Campo F, Thille AW, Cabello B, Galia F, Margarit L, d'Ortho MP, Brochard L. A new classification for sleep analysis in critically ill patients. Sleep Med. 2012 Jan;13(1):7-14. doi: 10.1016/j.sleep.2011.07.012. Epub 2011 Dec 6. PMID 22153778
- [Background] Rochwerg B, Granton D, Wang DX, Helviz Y, Einav S, Frat JP, Mekontso-Dessap A, Schreiber A, Azoulay E, Mercat A, Demoule A, Lemiale V, Pesenti A, Riviello ED, Mauri T, Mancebo J, Brochard L, Burns K. High flow nasal cannula compared with conventional oxygen therapy for acute hypoxemic respiratory failure: a systematic review and meta-analysis. Intensive Care Med. 2019 May;45(5):563-572. doi: 10.1007/s00134-019-05590-5. Epub 2019 Mar 19. PMID 30888444
- [Background] Nishimura M. High-Flow Nasal Cannula Oxygen Therapy in Adults: Physiological Benefits, Indication, Clinical Benefits, and Adverse Effects. Respir Care. 2016 Apr;61(4):529-41. doi: 10.4187/respcare.04577. PMID 27016353
- [Background] Sklar MC, Dres M, Rittayamai N, West B, Grieco DL, Telias I, Junhasavasdikul D, Rauseo M, Pham T, Madotto F, Campbell C, Tullis E, Brochard L. High-flow nasal oxygen versus noninvasive ventilation in adult patients with cystic fibrosis: a randomized crossover physiological study. Ann Intensive Care. 2018 Sep 5;8(1):85. doi: 10.1186/s13613-018-0432-4. PMID 30187270
- [Background] Rittayamai N, Phuangchoei P, Tscheikuna J, Praphruetkit N, Brochard L. Effects of high-flow nasal cannula and non-invasive ventilation on inspiratory effort in hypercapnic patients with chronic obstructive pulmonary disease: a preliminary study. Ann Intensive Care. 2019 Oct 22;9(1):122. doi: 10.1186/s13613-019-0597-5. PMID 31641959
- [Background] Roca O, Riera J, Torres F, Masclans JR. High-flow oxygen therapy in acute respiratory failure. Respir Care. 2010 Apr;55(4):408-13. PMID 20406507
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908